CLINICAL TRIAL: NCT00832702
Title: Women's Ischemia Syndrome Evaluation (WISE) Coronary Vascular Dysfunction
Status: Active, not recruiting | Type: Observational
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); University of Florida (Other); University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Noel Bairey Merz, Director, Cedars-Sinai Medical Center
Other Study IDs: IRB# 14906; 5R01HL090957 (NIH)
Record Dates: First submitted 2009-01-28; First posted 2009-01-30 (Estimated); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Cardiovascular Disease
Keywords: Cardiac; MRI; Coronary Vascular Dysfunction
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample will be collected for future genetic studies to better understand heart artery disease by identifing genetic factors that contribute to heart artery disorders, and for extraction and creation of cell lines.
Oversight: Data Monitoring Committee: No | US Export: No

INTERVENTIONS:
Procedure: Cardiac MRI — CMRI provides unique clinical utilities including excellent soft tissue characterization and contrast, three-dimensionality, quantitation of blood flow, and overall superior temporal and spatial resolution to image vascular and myocardial abnormalities.

SUMMARY:
This research study is designed to investigate the approaches to noninvasive detection and assessment of coronary vascular dysfunction in women by comparing the testing results from the invasive standard care diagnostic procedure Angiogram and from the additional noninvasive diagnostic procedure CMR Imaging. The investigators want to specifically study 375 female patients who have signs or symptoms suggestive of heart disease but don't have obstructive coronary artery disease. Two study sites (Cedars-Sinai Medical Center and University of Florida) are recruiting participants.

The standard of care procedures include demographics, review of recent clinical symptoms, review of medications being taken, a physical exam, pre-angiogram blood collection, chest x-ray, ECG and heart angiogram. The research procedures for this study are the cold pressor testing, blood/urine collection, health questionnaire, the post-angiogram ECG and cardiac MRI.

Patients will be asked to undergo heart angiogram testing to test for abnormalities in their heart arteries. If the heart angiogram shows that the patients do not have blockages in major heart arteries, then the patients will have coronary flow reserve measurement test (as part of the heart angiogram) to determine whether the patients have abnormally functioning of the small heart arteries. This test will be performed by infusing the three drugs: adenosine, acetylcholine and nitroglycerin. The three drugs are naturally occurring substances and have been used for routine heart angiograms.

Cardiac Magnetic Resonance (CMR) imaging may help us more easily and non-invasively detect abnormalities in the inner layer of the heart muscle resulting from the abnormal function of the heart arteries. All the 375 participants will undergo baseline CMR imaging test and a subgroup of 200 participants will undergo a second CMR imaging test at their at least 1-year followup visit.

Patients will be followed up using phone questionnaires at 6 weeks, 6 months for 5 years, and than annually for 20 years thereafter. Other procedures in this study include obtaining informed consent, review of demographics, physical examination, ECG, blood and urine tests, clinical symptoms, medications, questionnaires, etc. The core laboratories include Blood, Lipoprotein, Chemistry Core Lab, Reproductive Hormone Core Lab, Inflammatory Marker Core Lab, Oxidative Stress Core Lab, and Angiographic Core Lab. Additionally, GCRC at Cedars Sinai will process, store and ship samples as needed/required.

DETAILED DESCRIPTION:
See Brief Summary above.

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic angina or anginal equivalent;
2. Aged 18 years or older;
3. No obstructive CAD at coronary angiography (performed within the previous 24 months).
4. Competent to give informed consent.

Exclusion Criteria:

1. Obstructive CAD ≥ 50% luminal diameter stenosis in ≥ 1 epicardial coronary artery,
2. Acute coronary syndrome (defined by the ACC/AHA criteria, Braunwald 2000),
3. Primary valvular heart disease clearly indicating the need for valve repair or replacement;
4. Patients with concurrent cardiogenic shock or requiring inotropic or intra-aortic balloon support;
5. Prior or planned percutaneous coronary intervention or CABG,
6. Acute MI;
7. Prior non-cardiac illness with an estimated life expectancy < 4 years;
8. Unable to give informed consent;
9. Chest pain with a non-ischemic etiology (e.g.,pericarditis, pneumonia, esophageal spasm);
10. Contraindications to CMRI (e.g., AICD, pacemaker, untreatable claustrophobia or known angio-edema).
11. Contraindications to adenosine or Regadenoson (Lexiscan)
12. Women with intermediate coronary stenoses (> 20% but < 50% luminal diameter stenosis assessed visually at the time of angiography) will undergo clinically indicated IVUS testing based on the judgment of the operator; those determined to have flow-obstructing stenosis will be excluded from the overall study.
13. Participation in a research study that conflicts with the current WISE study.
14. Women with coronary stenosis ≥ 50% in any epicardial coronary artery, assessed visually at the time of angiography, will not be included in the CRT subgroup.

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women undergoing clinically-ordered coronary angiography for suspected ischemia will be recruited. See the inclusion and exclusion criteria for details.
Sampling Method: Non-Probability Sample
Enrollment: 433 (Estimated)
Dates: Start 2008-09-17 (Actual); Primary Completion 2015-09-15 (Actual); Study Completion 2051-08-31 (Estimated)

PRIMARY OUTCOMES:
Abnormal cardiac magnetic resonance imaging (CMRI) | 30 years
  Subjects will be contacted at 6-week followup and then annually indefinitely.

SECONDARY OUTCOMES:
Resource utilization and costs | 30 years
  Annual costs will include cardiovascular hospitalizations, coronary revascularizations and angiography, outpatient testing, and visits to generalists, specialists, nurse practitioners/ physician's assistants, or community clinics.
Persistent Chest Pain Symptoms | 30 years
  Detailed information on chest pain symptoms will include the traditional angina questionnaire and the WISE female angina questionnaire
Quality of Life Outcomes | 30 years
  Quality of life and functional capacity will be collected using the standard instruments of SAQ and DASI

CONTACTS AND LOCATIONS:
Overall Officials: C. Noel Bairey Merz, MD, FACC, Principal Investigator — Cedars-Sinai Medical Center; Carl J Pepine, MD, MACC, Principal Investigator — University of Florida
Locations (2):
- United States (2):
  - Cedars-Sinai Barbra Streisand Women's Heart Center, Los Angeles, California
  - University of Florida, Gainesville, Florida

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Landes S, Aldiwani H, Thomson L, Wei J, Al-Badri A, Mehta PK, Pedram M, Motwani M, Cook-Weins G, Sopko G, Pepine CJ, Merz CNB, Dey D. Pericardial fat volume is related to endothelial-mediated coronary blood flow in women with suspected coronary microvascular dysfunction. A report from the Women's Ischemia Syndrome Evaluation-Coronary Vascular Dysfunction (WISE-CVD) study. Am Heart J Plus. 2024 Mar 7;40:100379. doi: 10.1016/j.ahjo.2024.100379. eCollection 2024 Apr. PMID 38586431
- [Derived] Jalnapurkar S, Landes S, Wei J, Mehta PK, Shufelt C, Minissian M, Pepine CJ, Handberg E, Cook-Wiens G, Sopko G, Bairey Merz CN. Coronary endothelial dysfunction appears to be a manifestation of a systemic process: A report from the Women's Ischemia Syndrome Evaluation - Coronary Vascular Dysfunction (WISE-CVD) study. PLoS One. 2021 Sep 27;16(9):e0257184. doi: 10.1371/journal.pone.0257184. eCollection 2021. PMID 34570768
- [Derived] AlBadri A, Wei J, Quesada O, Mehta PK, Xiao Y, Ko YA, Anderson RD, Petersen J, Azarbal B, Samuels B, Henry TD, Cook-Wiens G, Handberg EM, Van Eyk J, Pepine CJ, Bairey Merz CN. Coronary Vascular Function and Cardiomyocyte Injury: A Report From the WISE-CVD. Arterioscler Thromb Vasc Biol. 2020 Dec;40(12):3015-3021. doi: 10.1161/ATVBAHA.120.314260. Epub 2020 Oct 8. PMID 33028098
- [Derived] Wei J, Bakir M, Darounian N, Li Q, Landes S, Mehta PK, Shufelt CL, Handberg EM, Kelsey SF, Sopko G, Pepine CJ, Petersen JW, Berman DS, Thomson LEJ, Bairey Merz CN. Myocardial Scar Is Prevalent and Associated With Subclinical Myocardial Dysfunction in Women With Suspected Ischemia But No Obstructive Coronary Artery Disease: From the Women's Ischemia Syndrome Evaluation-Coronary Vascular Dysfunction Study. Circulation. 2018 Feb 20;137(8):874-876. doi: 10.1161/CIRCULATIONAHA.117.031999. No abstract available. PMID 29459474
- [Derived] Thomson LE, Wei J, Agarwal M, Haft-Baradaran A, Shufelt C, Mehta PK, Gill EB, Johnson BD, Kenkre T, Handberg EM, Li D, Sharif B, Berman DS, Petersen JW, Pepine CJ, Bairey Merz CN. Cardiac magnetic resonance myocardial perfusion reserve index is reduced in women with coronary microvascular dysfunction. A National Heart, Lung, and Blood Institute-sponsored study from the Women's Ischemia Syndrome Evaluation. Circ Cardiovasc Imaging. 2015 Apr;8(4):10.1161/CIRCIMAGING.114.002481 e002481. doi: 10.1161/CIRCIMAGING.114.002481. PMID 25801710
- [Derived] Wei J, Mehta PK, Johnson BD, Samuels B, Kar S, Anderson RD, Azarbal B, Petersen J, Sharaf B, Handberg E, Shufelt C, Kothawade K, Sopko G, Lerman A, Shaw L, Kelsey SF, Pepine CJ, Merz CN. Safety of coronary reactivity testing in women with no obstructive coronary artery disease: results from the NHLBI-sponsored WISE (Women's Ischemia Syndrome Evaluation) study. JACC Cardiovasc Interv. 2012 Jun;5(6):646-53. doi: 10.1016/j.jcin.2012.01.023. PMID 22721660